CLINICAL TRIAL: NCT01549262
Title: Clinical Validation of Embryo Culture and Selection by Morphokinetic Analysis; a Randomized Controlled Trial by Time-lapse System
Brief Title: Clinical Validation of Embryo Cinematography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Marcos Meseguer, Embryologist IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1009-C-088-IR
Record Dates: First submitted 2012-02-16; First posted 2012-03-09 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Embryo Diagnosis and Selection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Incubator (Active Comparator)
  Interventions: Device: Observe embryo development
- ESD Time-lapse Monitoring system (Experimental)
  Interventions: Device: Observe embryo development with "Unisense FertiliTech A/S" (EC Certificte DGM - 673)

INTERVENTIONS:
Device: Observe embryo development with "Unisense FertiliTech A/S" (EC Certificte DGM - 673) — Observation of exact timing of embryo cleavages together with other morphology dynamics parameters.
  Arms: ESD Time-lapse Monitoring system
Device: Observe embryo development — Observe embryo development in the traditional manner
  Arms: Standard Incubator

SUMMARY:
The purpose of this study is to determine whether the multivariable model for embryo selection (Meseguer et al. 2012) together with undisturbed controlled conditions obtained by a time-lapse incubator system is effective in improving ongoing pregnancy rate in comparison with standard incubator and an embryo selection process based exclusively in morphology.

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing assisted reproduction with ICSI, first or second cycle
* 20 to 38 yers old
* BMI (18-25)
* No endometriosis,
* > 6 Metaphse II oocytes
* Basal FSH < 12 UI
* AMH > 7pmol/L

Exclusion Criteria:

* Hydrosalpinx
* Recurrent pregnancy loss
* Severe male factor

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 843 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Ongoing Pregnancy Rate | confirmed 16-18 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Valencia, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Insua MF, Cobo AC, Larreategui Z, Ferrando M, Serra V, Meseguer M. Obstetric and perinatal outcomes of pregnancies conceived with embryos cultured in a time-lapse monitoring system. Fertil Steril. 2017 Sep;108(3):498-504. doi: 10.1016/j.fertnstert.2017.06.031. PMID 28865550
- [Derived] Rubio I, Galan A, Larreategui Z, Ayerdi F, Bellver J, Herrero J, Meseguer M. Clinical validation of embryo culture and selection by morphokinetic analysis: a randomized, controlled trial of the EmbryoScope. Fertil Steril. 2014 Nov;102(5):1287-1294.e5. doi: 10.1016/j.fertnstert.2014.07.738. Epub 2014 Sep 11. PMID 25217875